CLINICAL TRIAL: NCT00454675
Title: Pulmonary Function Changes in 10 Pack Year Smokers With Chronic Bronchitis
Status: Completed | Type: Observational
Sponsor: Westside Family Medical Center, P.C. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Gary E. Ruoff, M.D., Westside Family Medical Center, P.C.
Other Study IDs: COPD-2006-01
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Bronchitis; COPD
Keywords: Smokers; Chronic Bronchitis; Pulmonary Function Test Abnormalities; COPD
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

SUMMARY:
To determine whether an average population of males and females who smoke 10 pack years or more of cigarettes in a primary care setting with chronic bronchitis has already developed significant changes on pulmonary function testing.

DETAILED DESCRIPTION:
The incident of COPD is dramatically increasing while other chronic disease states are decreasing in the US population. Smoking cigarettes is the leading risk factor for COPD. Smokers with chronic bronchitis may show early or late changes of COPD on pulmonary function tests. It is imperative that we define this patient population to determine whether early intervention will alter pulmonary function over the years.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign a written informed consent.
2. Enrollment population would include males and females 40 years of age to 80 years of age.
3. Current history or past history of smoking at least 10 pack years of cigarettes.
4. Patients to satisfy the diagnosis of chronic bronchitis.
5. Non-smokers will be allowed in the control group

Exclusion Criteria:

1. Chronic infections such as TB or other infections of the lungs.
2. Collagen diseases such as rheumatoid arthritis or lupus which affect the lungs.
3. Any previous lung diseases such as pneumoconiosis.
4. Previous accidents or surgery which would involve the lungs or the ribcage.
5. Maintenance medications used for asthma or COPD such as long acting bronchodilators or inhaled corticosteroids.
6. Asthma patients or other patients with allergies that may affect pulmonary function test will be excluded.
7. Any medical condition in the opinion of the investigator that would make the subject unsuitable for enrollment.
8. Pregnant woman will not be allowed
9. Current participation in a research study or within the last 30 days.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Ruoff, MD, Principal Investigator — Westside Family Medical Center, P.C.
Locations (1):
- Westside Family Medical Center, P.C., Kalamazoo, Michigan, United States